CLINICAL TRIAL: NCT04342624
Title: Effects of Cinnamon Spice on Glucose, Insulin, GI Hormone and Microbiome in Obese Individuals With Pre-Diabetes
Brief Title: Investigation of Cinnamon Spice on Glucose Tolerance in Subjects With Pre-diabetes
Acronym: CINNII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 19-002074
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes; Blood Glucose, High
Keywords: glucose; cinnamon; pre-diabetes; microbiome
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon (Experimental): Consume 4g of cinnamon capsules daily. Will be randomized, double blind, cross-over to other arm after.
  Interventions: Dietary Supplement: Cinnamon
- Placebo (Placebo Comparator): Consume 4g of placebo daily. Will be randomized, double blind, cross-over to other arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cinnamon — Cinnamon supplement
  Arms: Cinnamon
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine whether the effectiveness of cinnamon spice capsules vs. placebo capsules on glucose tolerance in prediabetic subjects who are overweight or obese.

DETAILED DESCRIPTION:
Participants will be asked to take cinnamon spice or placebo capsules daily with breakfast and dinner (2 weeks of cinnamon, 2 weeks of placebo). The placebo capsule is a study product that looks like the cinnamon capsules, but contains no active ingredients. The amount of cinnamon will be 4 grams per day. 2 grams will be taken at breakfast and dinner. Timed blood collections over a three-hour period will be used to measure how cinnamon spice affects glucose metabolism/insulin sensitivity in human subjects. Everyone who participates in the study will receive each treatment in random order. In this way, everyone will receive cinnamon spice capsules and placebo.

In a crossover study design subjects will consume either cinnamon or placebo with foods and before bed for 28 days. The placebo capsule is a study product that looks like the cinnamon capsules, but contains no active ingredients. The participants will also be asked to undergo an oral glucose tolerance test 4 times (on separate days) before and after the first and second cinnamon/placebo consumption. Subjects will take 3 capsules of cinnamon or placebo (total 2 g) with the glucose drink (75 g). Timed blood collections over a three-hour period will be used to measure how cinnamon spice affects glucose metabolism/insulin sensitivity in human subject. Continuous glucose monitoring will performed through the entire study for each subject. The microbiome will also be examined at the beginning and end of each 28 day phase (0-4 weeks and 6-10weeks). Subjects will consume a brown-beige diet during the study to exclude the effects of other polyphenol-rich foods. We will enroll twenty subjects >= 20 years of age, overweight/obese (BMI 25 to 35 kg/ m2) with fasting blood sugar between 100 and 126 mg/dl or HbA1c >=5.7% and <= 6.5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adults age >=20 years' old
* Typically consume low fiber/polyphenol diet (beige diet see below)
* Overweight/obese individuals with a BMI of 25 to 40 kg/m2 and HbA1c >=5.6% and <= 6.5%.
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* Any subjects with cinnamon intolerance
* Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Any subject currently taking blood thinning medications such as Warfarin or Coumadin
* Any history of gastrointestinal disease or surgery except for appendectomy or cholecystectomy.
* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement, which interfere with the absorption of polyphenols.
* History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP >95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history.
* Pregnant or breastfeeding
* Currently uses tobacco products.
* Currently has an alcohol intake >= 20 g ⁄ day;
* Currently has a coffee intake >= 3 cups ⁄ day;
* Allergy or sensitivity to cinnamon. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive history of cinnamon ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
* Is unable or unwilling to comply with the study protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose control using glucose tolerance test | 3 hours
  To determine the effect of cinnamon on glucose tolerance acutely after 75g glucose intake in pre-diabetic overweight/obese individuals
Blood glucose control with continuous glucose monitoring. | 4 weeks
  To determine the effect of cinnamon on glucose tolerance for 4 weeks in pre-diabetic overweight/obese individuals
Mircobiome effects of cinnamon through stool sample collection | 4 weeks
  To determine the effects of cinnamon on gut microbiota, short chain fatty acids, gut hormones GLP-1, GIP,glucagon and metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — UCLA Professor of Medicine
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Zelicha H, Yang J, Henning SM, Huang J, Lee RP, Thames G, Livingston EH, Heber D, Li Z. Effect of cinnamon spice on continuously monitored glycemic response in adults with prediabetes: a 4-week randomized controlled crossover trial. Am J Clin Nutr. 2024 Mar;119(3):649-657. doi: 10.1016/j.ajcnut.2024.01.008. Epub 2024 Jan 26. PMID 38290699